CLINICAL TRIAL: NCT06599190
Title: Effect Of Abdominal Hypopressive Training On Stress Urinary IncontinenceIn Female Athletes
Brief Title: Effect Of Abdominal Hypopressive Training On Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Badr University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Saeed Mohamed, lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004947
Record Dates: First submitted 2024-08-18; First posted 2024-09-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Female Stress Urinary Incontinence
Keywords: stress incontinence, and female athelete
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: They will be randomly distributed into 2 groups equal in numbers:
  Group (A) (Control group) consists of 25 female athletes. They will receive nutritional instructions and pelvic floor muscle exercises three sessions/week for 3 months.
  Group (B) (Study group) consists of 25 female athletes. They will receive the same treatment for the control group and abdominal hypopressive exercises three sessions/week of 30 mins per week for 3 months.
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Control group) (Active Comparator): consists of 25 female athletes. They will receive nutritional instructions and pelvic floor muscle exercises three sessions/week for 3 months.
  Interventions: Other: pelvic floor exercises, nutritional instructions
- Group (B) (Study group) (Experimental): consists of 25 female athletes. They will receive the same treatment for the control group and abdominal hypopressive exercises three sessions/week of 30 mins per week for 3 months.
  Interventions: Other: abdominal hypopressive exercises, pelvic floor exercises, nutritional instructions

INTERVENTIONS:
Other: pelvic floor exercises, nutritional instructions — They will receive nutritional instructions and pelvic floor muscle exercises three sessions/week for 3 months.
  Arms: Group (A) (Control group)
Other: abdominal hypopressive exercises, pelvic floor exercises, nutritional instructions — consists of 25 female athletes. They will receive the same treatment for the control group and abdominal hypopressive exercises three sessions/week of 30 mins per week for 3 months.
  Arms: Group (B) (Study group)

SUMMARY:
Fifty female athletes suffering from stress incontinence (SUI) will participate in this study. They will be selected from El Zohour Club, New Cairo City.

DETAILED DESCRIPTION:
They will be randomly distributed into 2 groups equal in numbers:

Group (A) (Control group) consists of 25 female athletes. They will receive nutritional instructions and pelvic floor muscle exercises three sessions/week for 3 months.

Group (B) (Study group) consists of 25 female athletes. They will receive the same treatment for the control group and abdominal hypopressive exercises three sessions/week of 30 mins per week for 3 months.

Before data collection, the purpose and procedures will be fully explained to the females. Informed consent will be obtained from each female. Each female will be evaluated following a standard protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Female athletes suffering from SUI.
2. They will be diagnosed with SUI using bladder stress test.
3. Their ages will range from 14-18 years old.
4. Their body mass index (BMI) will range from 18.5-24.9 kg/m2.
5. They are single females.

Exclusion Criteria:

The female athlete will be excluded if they had:

1. Urinary tract infection.
2. Family history of genito-urinary tract cancer.
3. Diabetes mellitus.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Assessment of urine loss | 24 hours pad test for12 weeks
  Pad testing will be used to quantify the volume of urine loss by weighing an absorbent pad before and after some type of leakage provocation. The test will start with weighting clean empty pad in grams. Then, it will be used until next time and weighted again. The weight of the used pad will be subtracted from the weight of the empty pad so the net result will determine the amount of leakage.
assesment of pelvic floor muscle contraction and tonning | 12 weeks
  The measurements will be taken in crock-lying position with a full bladder, neutral lumbar spine. The ultrasound transducer will be inserted transversely directly superior to the symphysis pubis, probe is tilted 60 degrees from vertical (Arab, 2010). Every female will perform 3 maximal PFM contractions so that displacement of the bladder wall, because of a PFM contraction, could be measured.

SECONDARY OUTCOMES:
Assessment of symptoms and health related quality of life | 12 weeks
  The ICIQ-SF will be used in assessment of each female in both groups. It is used to measure severity and impact of UI on the quality of life in women. The ICIQ-SF is formed of six items of which four main items ask for rating of UI symptoms in the past 4 weeks. A score of zero means no leakage of urine and no affection on quality of life. (Question 1): quantifies the frequency of urinary leaking, (question 2): evaluates the amount of leaking and (question 3): how much the urinary incontinence interferes with everyday life (Hilton and Robinson, 2011). The scores for items 3, 4 and 5 are taken for the final ICIQ-SF score. Items 1 and 2 are demographic and the final item is a self-diagnostic item for the type of UI. ICIQ- SF (range 0-21) is given four scoring categories: slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21).

CONTACTS AND LOCATIONS:
Overall Officials: Abeer ElDeeb, Professor, Study Chair — professor doctor
Locations (1):
- El Zohour Club, New Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
not sharing